CLINICAL TRIAL: NCT03834181
Title: Evaluation of a Telemedicine System for Patients Carried for Bariatric Surgery
Acronym: Bartélémis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-003
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Bariatric Surgery Candidate
Keywords: Connected devices; Telemetry; Obesity surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring evaluation (Experimental): Monitoring evaluation by connected devices: Wristband activity tracker "Garmin Vivosmart® 3", "Fora® Scale 550", "Terraillon® Tensioscreen", Pulse oximeter "Nonin® 3230", thermometer "Fora® IR20b"
  Interventions: Device: Monitoring evaluation by connected devices: Wristband activity tracker "Garmin Vivosmart® 3", "Fora® Scale 550", "Terraillon® Tensioscreen", Pulse oximeter "Nonin® 3230", thermometer "Fora® IR20b"

INTERVENTIONS:
Device: Monitoring evaluation by connected devices: Wristband activity tracker "Garmin Vivosmart® 3", "Fora® Scale 550", "Terraillon® Tensioscreen", Pulse oximeter "Nonin® 3230", thermometer "Fora® IR20b" — All patients will be monitored before and after the bariatric surgery:
  * During the preoperative preparation phase: weight, exercise, blood pressure and heart rate
  * In the immediate post operative period: continuous monitoring of the heart rate with a telemetry system
  * Prolonged follow-up: weight, exercise, blood pressure and heart rate

SUMMARY:
This study is intended to study the feasibility of a telemedicine system to monitor and control certain vital parameters before and after surgery for obesity. During the preoperative preparation phase, weight, exercise, blood pressure and heart rate are recorded and transmitted to the patient's surgeon. In the immediate post operative period, the heart rate is a sensitive and reliable indicator of the occurrence of a complication. A telemetry system will allow rapid home return, continuous monitoring and early warning in the event of a problem. Prolonged follow-up identical to that started preoperatively should allow improvement and better control of weight loss by monitoring especially physical exercise.

DETAILED DESCRIPTION:
The evolution of the health system requires a rationalization of the supply of care and the care of patients. It has allowed the evolution and generalization of ambulatory surgery for certain pathologies. For other pathologies, a hospital stay is still desirable with a tendency to decrease the length of stay. Thanks to the telemedicine platforms, specialized medical monitoring can be extended pre- and post-operatively to ensure good patient preparation and quality secure follow-up.

Early return to home is an essential parameter in optimizing the distribution of hospital resources. Several studies have shown improved clinical outcomes, fewer complications, more beds available, and lower hospital costs. The development of outpatient surgery has enabled the establishment of systems allowing a return home in secure conditions. Early return home is also a wish of the patient. He becomes an actor of his own health. Obesity surgery is an exemplary specialty for the care of patients. The ideal course of care is perfectly codified both preoperatively and postoperatively. Nevertheless, this ideal care path is not always respected especially in structures too small to offer a real integrated multidisciplinary follow-up. Pre- and postoperative management solutions on the Internet exist but require a voluntary and active adherence of the patient. They allow a stronger involvement of the patient in his approach, they are nascent and integrate no connected solution for automated monitoring of the patient. Telemedicine can now allow continuous monitoring without the need for face-to-face interaction. The automatic collection of the physical activity and the heart rate makes it possible to guarantee the involvement of the patient in his preparation. After the intervention, the monitoring of the occurrence of complications can be delegated to connected objects with alert transmission according to parameters defined in advance. In particular, the heart rate is a sensitive indicator and will be followed by two sensors (activity bracelet and pulse oximeter). These complications occur mainly in the 15 days following the intervention, they are rare in immediate postoperative. The hospital stay is no longer necessary for a simple surveillance. In case of receipt of an alert, the surgeon contacts the patient to check his state of health. An adapted action is then engaged.

The late postoperative follow-up throughout this document corresponds to the phase following the immediate postoperative phase. This late postoperative follow-up can be improved with the support of telemonitoring (activity, change in weight.) The addition of connected devices allows a stronger and faster interaction between the patient and his doctors, providing close monitoring and appropriate support.

The study focuses on assessing the reliability of a remote monitoring system. The implementation of this remote monitoring system is subordinated to the reliability of the data transmissions between the connected objects and the remote site which receives the data, interprets them and generates the alerts.

The motivation of the patient is appreciated by the acceptance of connected objects.

During this study, the remote monitoring system is offered in addition to the usual care. The usual care does not change and is not impaired. This study concerns only one group of patients, there is no control group since the investigators seek to validate the reliability of remote surveillance.

ELIGIBILITY:
Inclusion Criteria:

1. Patient (s) applying for bariatric surgery
2. Patient aged 18 to 65
3. Compliance with the High Authority of Health (HAS) criteria:

   * BMI> 40 without comorbidities
   * BMI> 35 with cardiovascular, metabolic, respiratory or rheumatic comorbidity,
   * Psychological follow-up well followed for 4 to 6 months
4. Patient with an ASA (American Society of Anesthesiologists) score less than or equal to 2
5. Patient able to receive and understand information about the study
6. Patient able to manipulate connected objects
7. Patient (e) affiliated to the French social security system
8. Patient who does not live in the white area of wireless telephone coverage.

Exclusion Criteria:

1. Patient unable to give informed consent
2. Patient unable to use the connected tools (Internet)
3. Patient whose general condition is not favorable to participation in the study
4. Patient presenting, in the opinion of the investigator, a condition that may prevent participation in the procedures provided for in the study
5. Patient in exclusion period (determined by previous or current study)
6. Patient under the protection of justice
7. Patient under guardianship or trusteeship
8. Patient with epilepsy
9. Patient who is sensitive to light flashes
10. Patient with deformity of the ear
11. Patient with bleeding ear

Exclusion Criteria :

1. Patient whose home is in a white GSM (Global System for Mobile Communications) zone or white zone in reception and 3G (third generation) transmission
2. Patient (e) not knowing how to use connected objects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Reliability of a remote monitoring system during treatment for bariatric surgery evaluated in days between two failures | From the inclusion to 6 months after the surgery
  The reliability of the system, corresponding to the average time between two failures, over the 9 months of study for each of the 30 patients. A failure is a momentary and abrupt loss of the ability of the system to transmit data.

SECONDARY OUTCOMES:
Patient acceptance of adding a telemonitoring device to their care evaluated in percentage of patients who signed a consent | Inclusion period of 4 months
  Acceptance is the ratio of the number of patients who signed the consent to the number of total patients to whom the study was presented as a percentage.
Relevance of the data received from each connected object (activity bracelet, scales, blood pressure monitor, thermometer and pulse oximeter) evaluated in percentage of data sent and verified | Study duration of 18 months
  The relevance of the data corresponds to the number of data sent and verified, using the alert system, of each of the connected objects (activity bracelet, scales, blood pressure monitor, thermometer and pulse oximeter) the number of data sent by the system over the entire duration of the study (activity bracelet, scale, tensiometer) or the entire immediate postoperative period (thermometer, pulse oximeter), in percentage.
Durability of the data over a defined period evaluated in number of connections. | From the inclusion to 6 months after the surgery
  The durability of the data corresponds to the number of connections interrupted or lost in a duration of more than 90 minutes per patient
Ratio of the number of patients who performed all the prescribed autonomic measures requested on the total number of patients included in the study | Study duration of 18 months
  Ratio of the number of patients who performed all the prescribed autonomic measures requested on the total number of patients included in the study, as a percentage. It will be evaluated by age categories (18-24, 25-34, 35-44, 45-54, 54-65 years), sex (male and female) and obesity classes (35.00 ≤ BMI). ≤ 39.99 kg / m² and BMI ≥ 40.00 kg / m²)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Vix, MD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loots E, Sartorius B, Paruk IM, Clarke DL. The Successful Implementation of a Modified Enhanced Recovery After Surgery (ERAS) Program for Bariatric Surgery in a South African Teaching Hospital. Surg Laparosc Endosc Percutan Tech. 2018 Feb;28(1):26-29. doi: 10.1097/SLE.0000000000000488. PMID 29064879
- [Background] Lemanu DP, Singh PP, Berridge K, Burr M, Birch C, Babor R, MacCormick AD, Arroll B, Hill AG. Randomized clinical trial of enhanced recovery versus standard care after laparoscopic sleeve gastrectomy. Br J Surg. 2013 Mar;100(4):482-9. doi: 10.1002/bjs.9026. Epub 2013 Jan 21. PMID 23339040
- [Background] Jonsson A, Lin E, Patel L, Patel AD, Stetler JL, Prayor-Patterson H, Singh A, Srinivasan JK, Sweeney JF, Davis SS Jr. Barriers to Enhanced Recovery after Surgery after Laparoscopic Sleeve Gastrectomy. J Am Coll Surg. 2018 Apr;226(4):605-613. doi: 10.1016/j.jamcollsurg.2017.12.028. Epub 2018 Jan 5. PMID 29309941
- [Background] Aman MW, Stem M, Schweitzer MA, Magnuson TH, Lidor AO. Early hospital readmission after bariatric surgery. Surg Endosc. 2016 Jun;30(6):2231-8. doi: 10.1007/s00464-015-4483-4. Epub 2015 Oct 19. PMID 26482158
- [Background] Kampmeijer R, Pavlova M, Tambor M, Golinowska S, Groot W. The use of e-health and m-health tools in health promotion and primary prevention among older adults: a systematic literature review. BMC Health Serv Res. 2016 Sep 5;16 Suppl 5(Suppl 5):290. doi: 10.1186/s12913-016-1522-3. PMID 27608677
- [Background] Wang Y, Xue H, Huang Y, Huang L, Zhang D. A Systematic Review of Application and Effectiveness of mHealth Interventions for Obesity and Diabetes Treatment and Self-Management. Adv Nutr. 2017 May 15;8(3):449-462. doi: 10.3945/an.116.014100. Print 2017 May. PMID 28507010
- [Background] Chen SY, Stem M, Schweitzer MA, Magnuson TH, Lidor AO. Assessment of postdischarge complications after bariatric surgery: A National Surgical Quality Improvement Program analysis. Surgery. 2015 Sep;158(3):777-86. doi: 10.1016/j.surg.2015.04.028. Epub 2015 Jun 19. PMID 26096563
- [Background] Montravers P, Augustin P, Zappella N, Dufour G, Arapis K, Chosidow D, Fournier P, Ribeiro-Parienti L, Marmuse JP, Desmard M. Diagnosis and management of the postoperative surgical and medical complications of bariatric surgery. Anaesth Crit Care Pain Med. 2015 Feb;34(1):45-52. doi: 10.1016/j.accpm.2014.06.002. Epub 2015 Mar 5. PMID 25829315